CLINICAL TRIAL: NCT02467985
Title: FIGARO : A Double-blinded RCT to Reduce Referred Pain in the Shoulder Following a Laparoscopic Gynecological Surgery
Brief Title: A Trial to Reduce Referred Pain in the Shoulder Following a Laparoscopic Gynecological Surgery
Acronym: FIGARO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, full professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-1042
Record Dates: First submitted 2015-05-11; First posted 2015-06-10 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Surgery
Keywords: gynecological laparoscopic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- intervention (Experimental): Flow of insufflation will be set to 2-3L / min. After the intervention, the CO2 insufflation is discontinued, accessories trocars are removed under direct vision and the incisions the sites of these trocars will be closed. Patients will be placed in the Trendelenburg position 30 degrees, head tilted down. The umbilical trocar is opened. Suction is inserted into the trocar, taking care to stay inside the jacket of the trocar. Active suction gas will during lung recruitment. This maneuver will be performed by the anesthesiologist who applies 5 subsequent forced breaths, up to 40 cm H2O pressure, taking care to maintain the insufflation last 5 sec. Once completed, the suction will be removed, the laparoscope is inserted into the trocar to verify the absence of trauma to underlying structures.
  Interventions: Procedure: FIGARO

INTERVENTIONS:
Procedure: FIGARO — flow of insufflation set to 2-3L / min. Once the intervention is complete, the CO2 insufflation is discontinued, accessories trocars are removed under direct vision and the incisions the sites of these trocars will be closed with or without fascial closure according to the standard display. Patients will be placed in the Trendelenburg position 30 degrees, head tilted down. The umbilical trocar is opened. A suction is inserted into the trocar, taking care to stay inside the jacket of the trocar. Active suction gas will during lung recruitment. This maneuver will be performed by the anesthesiologist who apply 5 subsequent forced breaths, up to 40 cm H2O pressure, taking care to maintain the insufflation last 5 seconds. Once completed, the suction will be removed, the laparoscope is inserted into the trocar to verify the absence of trauma to underlying structures. The patient will be given to neutral at the end of the procedure.
  Arms: intervention

SUMMARY:
Patients undergoing laparoscopic surgery suffer in 30-85% of cases of referred pain in the shoulder in the first days following their intervention. Pain can be disabling and may even delay the discharge of patients. Several techniques have been proposed to reduce this problem. Promising strategies include the reduction of CO2 insufflation flow, lung recruitment maneuvers and active aspiration of intraperitoneal air at the end of surgical procedure to force gas discharge. The investigators wish to perform a randomized controlled trial with 160 women, who will assess the effect of a combined approach, combining for the first time lung recruitment maneuvers and aspiration of pneumoperitoneum in the Trendelenburg position at the end of surgery and flow of insufflation reduces carbon dioxide (CO2) forming the pneumoperitoneum during surgery, on the intensity of shoulder pain postoperatively. In the control group the evacuation of the pneumoperitoneum will be done by opening the trocars and external abdominal pressure at the end of surgery. No study to our knowledge has tested the active aspiration maneuvers gas after laparoscopic surgery in gynecology. The study will be preceded by a pilot study in 15 participants, who will be assigned to the control group to determine the basic rate of referred pain in the shoulder in our people and improve test management.

ELIGIBILITY:
Inclusion Criteria:

* women, 18-65 years
* physical ASA score 1-2
* Elective laparoscopic surgery for benign cause
* patients who have been informed of the study and has agreed to sign the ICF

Exclusion Criteria:

* physical ASA score 3-4
* pregnant women
* chronic pain syndrome or preoperative pain syndrome
* narcotics consumption, chronic preoperative analgesia
* alcohol or drug dependence
* inability to provide telephone follow up at 48 hours
* laparoscopy not possible at the umbilical level.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
shoulder pain | 48 hours
  questionnaire

SECONDARY OUTCOMES:
The impact of referred pain in the shoulder | 48 hours
  questionnaire
The intensity of abdominal pain Postoperatively | 48 hours
  questionnaire
The incidence of postoperative nausea | 48 hours
  questionnaire
The quality of life | 48 hours
  questionnaire
Theincidence of abdominal pain Postoperatively | 48 hours
  questionnaire
The incidence of postoperative vomiting | 48 hours
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada